CLINICAL TRIAL: NCT04748211
Title: Effect of Infraclavicular and Interscalen Block on Oxygenitaon of the Forearm : Randomized Controlled Study.
Brief Title: Effect of Infraclavicular and Interscalen Block on Oxygenitaon of the Forearm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, OZCAN PISKIN, MD, associate professor, Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-116-06/12
Record Dates: First submitted 2020-12-13; First posted 2021-02-10 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Upper Extremity Fracture

STUDY DESIGN:
Intervention Model Description: The study will be a two-arm parallel assignment. One group will receive infraclavicular block and the other will receive interscalen block
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infraclavicular Block (Experimental): Group I received USG and neurostimulator guided infraclavicular block, 10 ml 2% lidocain and 10 ml 0.05% marcaine was administered for local anetshesia. After the block was administered MAP, HR, TAV, BAD, BAA, BF, PI and rSO 2 values were measured and recorded at the 10th, 20th, and 30th minutes.
  Interventions: Procedure: Infraclavicular Block
- Interscalen Block (Experimental): Group II received USG and neurostimulator guided interscalen block. 10 ml 2% lidocain and 10 ml 0.05% marcaine was administered for local anetshesia. After the block was administered MAP, HR, TAV, BAD, BAA, BF, PI and rSO 2 values were measured and recorded at the 10th, 20th, and 30th minutes.
  Interventions: Procedure: Interscalen Block

INTERVENTIONS:
Procedure: Infraclavicular Block — USI and neurostimulator guided infraclavicular block, 10 ml 2% lidocain and 10 ml 0.05% marcaine was administered for local anetshesia. After the block was administered MAP, HR, TAV, BAD, BAA, BF, PI and rSO 2 values were measured and recorded at the 10th, 20th, and 30th minutes.
  Arms: Infraclavicular Block
Procedure: Interscalen Block — USI and neurostimulator guided interscalen block, 10 ml 2% lidocain and 10 ml 0.05% marcaine was administered for local anetshesia. After the block was administered MAP, HR, TAV, BAD, BAA, BF, PI and rSO 2 values were measured and recorded at the 10th, 20th, and 30th minutes.
  Arms: Interscalen Block

SUMMARY:
to research the oxygenitaon effects of infraclavicular and interscalene blocks on the forearm.

DETAILED DESCRIPTION:
To research the oxygenation effects of infraclavicular and interscalen blocks on the forearm by comparing the blood flow (BF) values using the USG, Perfusion index (PI) and Near infrared spectroscopy (NIRS) values using the massimo device.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18-65
* ASA Score I-III
* undergoing elective or emergency arm, elbow and forearm surgery

Exclusion Criteria:

* Patient's refusal for Brachial Plexus Blockage
* Patients who had any neurological disorders preventing the evaluation of the sensory block in the upper extremity,
* Infection in the area to be blocked with ICB or ISB,
* Non-cooperated patients
* Patients with coagulopathy,
* Morbidly obese patients
* Patients with diabetes mellitus
* Patients with hypertension
* Patients with peripheral artery disease
* Patients with allergy to the drugsto be used
* Patients who had trauma in the area scheduled for the block
* Paitens who had deterioration of anatomical integrity because of previous surgery
* Pregnant women
* Patients whose block failed

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
oxygenation of the forearm | during the procedure three times
  to compare the oxygenation of the forearm by measuring perfusion index device

CONTACTS AND LOCATIONS:
Overall Officials: Eren Açıkgöz, M.D., Principal Investigator — Bulent Ecevit University
Locations (1):
- Zonguldak Bulent Ecevit University, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No